CLINICAL TRIAL: NCT06751420
Title: Exploring Variants of Circle of Willis Through 3 Dimensional Time-of-Flight Magnetic Resonance Angiography Imaging: A Retrospective Cross Section Study
Brief Title: Circle of Willis Variants in Nepali Population Evaluated in TOF MR Angiography
Acronym: COW
Status: Completed | Type: Observational
Sponsor: Grande International Hospital, Nepal (Other)
Responsible Party: Principal Investigator, PRAJWAL DAHAL, Principal Investigator, Grande International Hospital, Nepal
Other Study IDs: 11/2024; GIH (Other: Grande International Hospital)
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Circle of Willis; Aneurysm, Congenital, Ruptured
Keywords: Circle of Willis; Time Of Flight Magnetic Resonance Angiogram; Brain
MeSH Terms: conditions — Aneurysm; Rupture | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — Magnetic Resonance Imaging Time Of Flight Angiography

SUMMARY:
The brain, though it constitutes only 2% of total body weight, receives 20% of the cardiac output. Blood supply to the brain comes from two major pairs of arteries: the anterior carotid arteries and the posterior vertebral arteries, which form an important collateral network. This network ensures that blood flow is maintained even if one of the arteries is obstructed. In 1664, Sir Thomas Willis first described this system, which was later named the "Circle of Willis" (COW) after him. Normally, there is little blood mixing between the branches of the circle, but during blockages in the main arteries, these collaterals can activate to maintain cerebral perfusion. The COW consists of an anterior and posterior portion. The anterior portion, supplied by the carotid arteries and their branches, and the posterior portion, formed by the vertebrobasilar system, provide critical blood flow to the brain. The key arteries involved in the COW include the internal carotid arteries (ICAs), anterior cerebral arteries (ACAs), anterior communicating artery (ACom), posterior cerebral arteries (PCAs), basilar artery (BA), and posterior communicating arteries (PComs). Anatomical variations in the COW are common, with a complete arterial circle being rare. Studies have documented a range of normal variants of the COW, which are likely to arise during vasculogenesis. Magnetic resonance imaging (MRI), using the non-invasive time of flight (TOF) technique, is a cost-effective and contrast-free method for visualizing the COW in three dimensions, making it preferable to conventional angiography.

The variants of COW and diameters of arteries of COW are of clinical importance given its critical role in brain blood supply. Understanding CoW variants can reveal predispositions to conditions like stroke and aneurysms. This research will provide prevalence data on CoW configurations, aiding diagnostic and treatment strategies for cerebrovascular diseases, and may offer insights into vascular development influences.

DETAILED DESCRIPTION:
A study from Nepal conducted by Sharma et al.(1) investigated anatomical variations of the Circle of Willis (CoW) in the Nepalese population using 3D Time-of-Flight Magnetic Resonance Angiography (TOF-MRA). Among 118 subjects, only 46.6% exhibited the typical CoW configuration, with the most common variation being the absence or hypoplasia of the posterior communicating artery (PCOM), particularly the right PCOM (13.6% of cases). The findings suggest that morphological variations in CoW are common in Nepal, similar to global studies. Notably, women were more likely to present variant configurations than men, though no age-related trends in CoW morphology were observed. A study similar to our was done by Kızılgöz et al.(2) in Turkish population. This study enrolled 867 patients who had undergone MR angiography (MRA) to assess the Circle of Willis (CoW). Using three-dimensional time-of-flight MRA images, the researchers re-evaluated vessel diameters across all CoW components and classified CoW variations. They also analyzed how vessel calibers and CoW integrity related to gender and age groups. The study had a higher proportion of female participants, with an average age of 48. Type A was the most frequent variation in both anterior (75.78%) and posterior (53.98%) circulations. In the anterior circulation, types G and H were also common, while types E and D were the second and third most frequent in the posterior CoW, respectively. Females generally had smaller calibers in both ICAs, both P1s, and the BA compared to males. In patients with a complete CoW, the diameters of the BA and both P1 segments were lower, while the left PCom diameter was significantly larger. There was a notable variation by sex and age in the distribution of complete, partially complete, and incomplete CoW configurations. These findings on vessel calibers in complete, partial, and incomplete CoWs suggest that further research is needed, and meta-analyses with other studies could provide insights into CoW morphology. A study from India by Naveen et al.(3) examined CoW configurations in a South Indian population using TOF-MRA on 300 subjects. They found that only 16.6% had a complete CoW, with the most frequent variation being hypoplasia or absence of PCOM, observed predominantly in the posterior circulation. Incomplete CoW configurations were more common in older adults, with significant differences between age and sex groups. These findings highlight the CoW's role as a collateral pathway and its potential impact on cerebrovascular health. In Norway, Hindenes et al.(4) studied CoW variants in a large population using 3D TOF-MRA. They identified 47 unique configurations, with the complete CoW variant found in only 11.9% of cases. The study revealed that missing posterior communicating arteries were most common and associated with older age, indicating reduced collateral capacity. No significant sex differences were noted. This study underscores the CoW's variability and the effect of aging on its structure, emphasizing the clinical significance of collateral pathways in cerebrovascular health. Another study done by Diljohn et al. in Trinidian population showed complete Circle of Willis (CoW) in 24.3% of participants, with a higher occurrence in younger individuals (≤45 years) and Afro-Trinidadians. No gender preference for a complete CoW was identified. The most frequent variations in the CoW were a hypoplastic anterior communicating artery (8.6%, n=13) and bilateral aplastic posterior communicating arteries (18.4%, n=28) in the anterior and posterior segments, respectively.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (18+ years) with high-quality, three-dimensional time-of-flight MR angiography (TOF-MRA) imaging that clearly visualizes the Circle of Willis (CoW) and is performed for neurological assessments, such as headache or transient ischemic attacks.

Exclusion Criteria:

* patients with incomplete or poor-quality imaging, prior neurosurgical interventions, or significant vascular pathologies (e.g., aneurysms, arteriovenous malformations, severe atherosclerosis) that could distort natural CoW anatomy. Additionally, images with motion artifacts and cases with missing essential demographic or clinical information are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of all gender and age 18 and above
Sampling Method: Non-Probability Sample
Enrollment: 383 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of different type of anterior and posterior circulation | 6 months
  Prevalence of different type of anterior and posterior circulation in Nepali population

CONTACTS AND LOCATIONS:
Overall Officials: PRAJWAL DAHAL, MD, Principal Investigator — Grande International Hospital
Locations (1):
- Tokha Road, Dhapasi, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No